CLINICAL TRIAL: NCT07187635
Title: The Guiding Value of Urinary Tumor DNA Testing in Repeat Transurethral Resection of Non-Muscle-Invasive Bladder Cancer: An Open-Label, Randomized Controlled, Multi-Center Clinical Study (Truce-LB01)
Brief Title: Guiding Value of Urinary Tumor DNA Testing in Repeat Transurethral Resection of Non-Muscle-Invasive Bladder Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Truce-LB01
Record Dates: First submitted 2025-09-11; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-07

CONDITIONS: Bladder Cancer; Liquid Biopsy; Repeat Transurethral Resection of Bladder Tumor
Keywords: bladder cancer; liquid biopsy; second transurethral resection of bladder tumor
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard re-TURBT (Active Comparator): Participants with NMIBC who have undergone initial TURBT will not receive utDNA testing and will undergo a second transurethral resection of bladder tumor (re-TURBT) within 2-6 weeks after the initial surgery, per guideline-based management.
  Interventions: Procedure: Second Transurethral Resection of Bladder Tumor (re-TURBT)
- utDNA-guided management (Experimental): Participants with NMIBC who have undergone initial TURBT will receive urine tumor DNA (utDNA) testing.
  If utDNA positive, they will undergo re-TURBT within 2-6 weeks after the initial surgery.
  If utDNA negative, re-TURBT will be omitted and patients will continue guideline-based adjuvant therapy/surveillance as per protocol.
  Interventions: Diagnostic Test: utDNA Testing (Urine Tumor DNA Detection)

INTERVENTIONS:
Procedure: Second Transurethral Resection of Bladder Tumor (re-TURBT) — Participants with NMIBC who have undergone initial TURBT will not receive utDNA testing and will undergo a second transurethral resection of bladder tumor (re-TURBT) within 2-6 weeks after the initial surgery, in accordance with current clinical guidelines.
  Arms: Standard re-TURBT
Diagnostic Test: utDNA Testing (Urine Tumor DNA Detection) — Participants with NMIBC who have undergone initial TURBT will receive urine tumor DNA (utDNA) testing.
  If utDNA is positive, the patient will undergo a second transurethral resection of bladder tumor (re-TURBT) within 2-6 weeks after the initial surgery.
  If utDNA is negative, re-TURBT will be omitted and patients will proceed to guideline-based adjuvant therapy or surveillance.
  Arms: utDNA-guided management

SUMMARY:
Non-muscle-invasive bladder cancer (NMIBC) accounts for approximately 75% of newly diagnosed bladder cancers and is characterized by a high risk of recurrence and progression. Current guidelines recommend that patients with stage T1 NMIBC undergo a second transurethral resection of bladder tumor (re-TURBT) within 2-6 weeks after the initial surgery to remove residual tumor, confirm staging, and obtain additional pathological information. However, the benefits of routine re-TURBT for all high-risk patients remain controversial, as many patients may not have residual disease, while the procedure carries surgical and anesthetic risks, physical and psychological burden, and additional healthcare costs.

Urine tumor DNA (utDNA) refers to DNA fragments shed by tumor cells into urine. It can be detected using molecular assays with high sensitivity and specificity, offering a non-invasive method for bladder cancer diagnosis and surveillance. Previous studies have shown that positive utDNA results after initial TURBT may be associated with residual disease and higher recurrence risk.

This multicenter, randomized controlled trial aims to evaluate whether utDNA testing can accurately identify NMIBC patients who are most likely to benefit from re-TURBT, thereby guiding the decision to perform the procedure. The goal is to optimize patient selection for re-TURBT, reduce unnecessary surgeries, and improve patient quality of life while maintaining oncologic safety.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for the study:

1. Male or female, aged 18 years or older.
2. Histologically confirmed non-muscle-invasive bladder tumor, with no evidence of muscle-invasive bladder cancer or metastatic disease.
3. Histologically confirmed urothelial carcinoma of the bladder or bladder tumor with urothelial carcinoma as the predominant component (>50%).
4. At least one of the following conditions:

   1. Incomplete initial transurethral resection of bladder tumor (TURBT) or suspected incomplete resection.
   2. Absence of detrusor muscle in the initial TURBT pathological specimen (except for low-grade Ta stage tumors or carcinoma in situ [CIS]).
   3. T1 stage tumor.
5. Willingness to provide a 50 mL urine sample between 2-6 weeks after the initial TURBT and prior to re-TURBT.
6. Willingness to provide tumor tissue samples for pathological examination.
7. Willingness to undergo genetic testing required for the trial.

Exclusion Criteria:

1. Contraindications to transurethral resection of bladder tumor (TURBT).
2. Concurrent malignancy of the upper urinary tract (ureter or renal pelvis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | Up to 24 months from randomization
  Time from randomization to the first documented event of bladder tumor recurrence (any grade), upper tract urothelial recurrence.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 24 months from randomization
  Time from initial TURBT to disease progression (development of muscle-invasive bladder cancer, distant metastasis).
Pathological outcomes of second transurethral resection (re-TURBT) | Perioperative (day of repeat TURBT)
  Proportion of patients with residual tumor, upstaging (higher T category at re-TURBT), or concomitant CIS among those undergoing repeat TURBT.

OTHER OUTCOMES:
Correlation Between utDNA Status and Clinical Outcomes | Up to 24 months from randomization
  Association of urine utDNA results with cystoscopy findings, imaging results, and re-TURBT pathology; evaluation of diagnostic performance (sensitivity, specificity, predictive values, AUC) and relation to recurrence/progression.

CONTACTS AND LOCATIONS:
Locations (1):
- The second hospital of Tianjin Medical University, Tianjin, China